CLINICAL TRIAL: NCT00274131
Title: Long-term Administration Study of SND 919 Tablets in Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 248.506
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

INTERVENTIONS:
Drug: Pramipexole 0.125 mg tablets
Drug: Pramipexole 0.5 mg tablets

SUMMARY:
To evaluate the efficacy and safety of long-term treatment with pramipexole tablets (BI Sifrol®) in Parkinson's disease (phase III study).

DETAILED DESCRIPTION:
The efficacy and safety of long-term treatment with pramipexole (BI Sifrol®) were evaluated in Parkinson disease patients in an open-label non-controlled design. The treatment was initiated at 0.125 mg bid (after breakfast and supper).

The dose was increased stepwise with due caution regarding the symptoms and safety of each patient, up to 1.5 mg tid (after each meal). The treatment period was set at 56 weeks, followed by a stepwise dosedecreasing period (maximum 4 weeks).

Study Hypothesis:

Comparison(s):

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of Parkinson's disease (including juvenile parkinsonism)

(1) Patients meeting all of the following inclusion criteria

1. Patients of at least 20 years of age
2. In- or outpatients of either sex.
3. Patients in any stage on the modified Hoehn and Yahr severity scale

Exclusion Criteria:

* Patients with psychiatric symptoms such as confusion, hallucination, delusion, excitement, delirium, and abnormal behaviour.
* Patients with subjective symptoms derived from orthostatic hypotension.
* Patients with hypotension (systolic blood pressure <100 mmHg)
* Patients with concomitant illness such as severe cardiac, renal, and hepatic disease
* Patients with a current or past history of epilepsy
* Pregnant, possibly pregnant, or lactating women
* Patients receiving any other investigational products or who have received any other investigational product within 6 months of the study.
* Patients who judged incompetent to give consent
* Others judged by the investigator or co-investigator to be ineligible as subjects.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170
Dates: Start 1998-12; Study Completion 2004-02

PRIMARY OUTCOMES:
UPDRS Part II (activities of daily living) total score UPDRS Part III (motor examination) total score

SECONDARY OUTCOMES:
UPDRS Part I (mentation, behaviour and mood) total score UPDRS Part IV (complications of therapy) total score UPDRS Part I-III total score UPDRS Part I-IV total score Modified Hoehn and Yahr scale score Global impression of efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Nippon Boehringer Ingelheim Co., Ltd.